CLINICAL TRIAL: NCT02935764
Title: Phase III Study of Fluorouracil, Leucovorin, and Irinotecan Regimen (FOLFIRI) Versus Irinotecan Monodrug as Second-line Treatment in Metastatic Colorectal Cancer Patients
Brief Title: FOLFIRI Versus Irinotecan as Second-line Treatment in Metastatic Colorectal Cancer Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Weijian Guo, Vice Director of Department of Medical Oncology, Clinical Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDZL-FCI
Record Dates: First submitted 2016-10-04; First posted 2016-10-17 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Irinotecan; Fluorouracil; Leucovorin

ARMS (2):
- FOLFIRI (Experimental): 5-fluorouracil,folinate combined with irinotecan
  Interventions: Drug: Irinotecan; Drug: 5-fluorouracil; Drug: Leucovorin
- IRINOTECAN (Active Comparator): irinotecan
  Interventions: Drug: Irinotecan

INTERVENTIONS:
Drug: Irinotecan — 180 mg/m2 iv gtt, d1
Drug: 5-fluorouracil — 5-FU 400mg/m2 iv, 2400mg/m2 civ 46h
  Other Names: 5-FU
  Arms: FOLFIRI
Drug: Leucovorin — 400mg/m2 iv gtt,d1
  Other Names: LV
  Arms: FOLFIRI

SUMMARY:
This study is designed to compare the efficacy and safety of FOLFIRI regimen with irinotecan monodrug in the treatment of advanced colorectal cancer patients in the second-line setting.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-70 years with histologically or cytologically confirmed advanced colorectal adenocarcinoma
* Eastern Cooperative Oncology Group performance status of 0 to 2
* life expectancy of ≥ 3 months
* patients who had failed first-line treatment with either XELOX (capecitabine combined with oxaliplatin) or FOLFOX (5-fluorouracil/leucovorin with oxaliplatin)
* at least one measurable disease lesion according to the Response Evaluation Criteria in Solid Tumors (RECIST 1.1) criteria
* have adequate bone marrow, hepatic, and renal function

Exclusion Criteria:

* patients with previous chronic inflammatory bowel disease, chronic diarrhea or recurrent bowel obstruction
* patients with symptomatic brain metastases
* active clinical severe infection
* previously received irinotecan
* dihydropyrimidine dehydrogenase (DPD) enzyme adequate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2016-10; Primary Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
progression free survival | 2 months

SECONDARY OUTCOMES:
overall survival | 6 months
overall response rate | 2 months
Number of Participants with Adverse Events | 2 months
quality of life questionnaire | 2 months

REFERENCES:
- [Derived] Zhang X, Duan R, Wang Y, Liu X, Zhang W, Zhu X, Chen Z, Shen W, He Y, Wang HQ, Huang M, Wang C, Zhang Z, Zhao X, Qiu L, Luo J, Sheng X, Guo W. FOLFIRI (folinic acid, fluorouracil, and irinotecan) increases not efficacy but toxicity compared with single-agent irinotecan as a second-line treatment in metastatic colorectal cancer patients: a randomized clinical trial. Ther Adv Med Oncol. 2022 Jan 13;14:17588359211068737. doi: 10.1177/17588359211068737. eCollection 2022. PMID 35069808